CLINICAL TRIAL: NCT00605995
Title: Add-on Simvastatin in Schizophrenia Trial
Acronym: ASSIST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was slower than anticipated by the investigators and the funding research foundation.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Stanley Medical Research Institute (Other); Sheba Medical Center (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5207; SMRI-05T-693 (Other: protocol)
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2012-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Randomized trial; Statin; Placebo
MeSH Terms: conditions — Schizophrenia | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): Simvastatin, 20 mg Tablet, given once daily. Dosage increased to 40 mg/day at the end of week 4 until endpoint.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo pill, similar in its appearance to Simvastatin, taken once daily for the duration of the trial.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — 20 mg taken orally once daily for the first 4 weeks. Dosage will be increased to 40 mg/day at the end of week 4.
  Other Names: Zocor

SUMMARY:
The overall purpose of this study is to determine whether the cholesterol-lowering drug simvastatin is effective in the treatment of symptoms of schizophrenia. The primary hypothesis is that patients with schizophrenia receiving add-on treatment with simvastatin will improve clinically (as measured mainly by symptom severity) compared with patients receiving placebo, and that this improvement will be accompanied by concomitant reduction in peripheral inflammatory markers.

DETAILED DESCRIPTION:
The identification of alternative therapies with the capacity to dampen inflammatory processes and reduce serum cholesterol takes on additional significance given independent concerns about heightened cardiovascular risk in schizophrenia patients, through exposure to antipsychotic drugs, increased cholesterol levels, metabolic syndrome and obesity, and smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Available for follow up during the study protocol
* DSM-IV schizophrenia
* Positive and Negative Syndrome Scale (PANSS) baseline score of ≥50
* Score of 3 or higher on the Severity of Illness scale of the Clinical Global Impression (CGI)
* Not completely refractory to antipsychotics: evidence for at least partial responsiveness to antipsychotic medication
* Evidence for current clinical stability
* Capacity to provide informed consent
* Provided informed consent
* Patients taking concomitant, non-investigational medications that are not listed in Exclusion Criteria #1
* Patients speaking Spanish or English
* Women using acceptable methods of birth control, including barrier method

Exclusion Criteria:

* Currently taking a statin OR any of the following:

  * Other lipid-lowering drug;
  * Anti-inflammatory drugs or aspirin;
  * Systemic antibiotic, anti-viral or anti-fungal drugs (within the past 4 weeks);
  * Potent inhibitors of the cytochrome P450 isoform 3A4 (CYP3A4);
  * Digoxin (Lanoxin®), nefazodone (Serzone®), niacin, cyclosporine (Neoral®, Sandimmune®), danazol, warfarin (Coumadin®), amiodarone, verapamil, Cordarone®, or Inderal®.
* Patients with known hypersensitivity to simvastatin or any other statin drug
* Active liver disease or unexplained persistent elevations of serum transaminases
* Renal insufficiency
* Serious or unstable medical condition that require close medical attention, such as cancer, unstable heart failure, uncontrolled hypertension/asthma/COPD
* Current drug use disorder (abuse/dependence)
* Pregnancy and lactation
* Psychiatric disorders other than schizophrenia or schizoaffective disorder requiring pharmacotherapy
* Suicidal or homicidal intent
* Severe cognitive impairment that might compromise competency to sign informed consent or the validity of the cognitive outcome measure
* Organic brain disorder, including epilepsy; mental retardation; or a medical condition whose pathology or treatment would likely alter the presentation or treatment of schizophrenia
* Current participation in another clinical trial
* Patients on more than 2 anti-psychotic medications (patients will not be tapered off effective medications for the purpose of participating in research)
* LDL cholesterol >100 mg/dL with known coronary hard disease. LDL cholesterol >130 mg/dl with 2 or more of the following risk factors: smoking; hypertension; low HDL cholesterol (<40 mg/dL); age >45 years (men) or age >55 years (women); family history of premature CHD (CHD in 1st degree relative male<55; female <65

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Positive and negative symptoms of schizophrenia | 12 weeks

SECONDARY OUTCOMES:
Serum inflammatory markers and cholesterol levels. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raz Gross, M.D., MPH, Principal Investigator — Columbia University
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel